CLINICAL TRIAL: NCT00652795
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Doxycycline 150 mg Tablet and Monodox 50 mg Capsule Administered as 1 x 150 mg Tablet or 3 x 50 mg Capsules in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study Doxycycline Tablets and Monodox Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 40074
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: bioequivalence; doxycycline monohydrate; fasting
MeSH Terms: conditions — Fasting | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received the Par product (Doxycycline Monohydrate) under fasting conditions.
  Interventions: Drug: Doxycycline Monohydrate
- B (Active Comparator): Subjects received the Oclassen's product (Monodox) Capsules under fasting conditions.
  Interventions: Drug: Monodox

INTERVENTIONS:
Drug: Doxycycline Monohydrate — Tablets, 150 mg, single-dose
  Other Names: Monodox
  Arms: A
Drug: Monodox — Capsules 50 mg (3 x 50 mg dose), single-dose
  Other Names: Doxycycline Monohydrate
  Arms: B

SUMMARY:
To compare the rate and extent of absorption of doxycycline tablet (Par) versus doxycycline capsule (Monodox)(Oclassen).

DETAILED DESCRIPTION:
To compare the rate and extent of absorption of doxycycline 150 mg tablet (test) versus Monodox 50 mg capsule (reference) administered as 1 x 50 mg tablet or 3 x 50 mg capsules under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential female, smoker or non-smokers
* 18 years of age and older
* Non-childbearing potential female subjects is defined as post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy with bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration
* Capable of consent

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication
* Clinically significant surgery within 4 weeks prior to the administration of the study medication
* Any clinically significant abnormality found during medical screening
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study
* Abnormal laboratory tests judged clinically significant
* Positive testing for hepatitis B, hepatitis C or HIV at screening
* ECG abnormalities or vital sign abnormalities at screening
* BMI greater than or equal to 30.0 kg/m2
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week
* History of drug abuse or use of illegal drugs: soft drugs (marijuana) within 3 months prior to the screening visit or hard drugs (cocaine, PCP, crack) within 1 year prior to the screening visit or positive urine drug screen at screening
* History of allergic reactions to heparin, doxycycline, or other related drugs
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication
* Use of an investigational drug or participation in an investigational study, within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption
* Difficulty to swallow study medication
* Smoking more than 25 cigarettes per day Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in the study A depot injection or an implant of any drug within 3 months prior to administration of study medication
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study)prior to the administration of the study medication (50 mL to 300 mL of whole blood within 30 days, 301 mL to 500 mL of whole blood within 45 days, or more than 500 mL of whole blood within 56 days prior to drug administration)
* History or presence of clinically significant gastro-oesophageal reflux, stomach ulcers, or indigestions
* History or presence of clinically significant severe renal or hepatic dysfunction
* History or presence of clinically significant myasthenia gravis
* Breast-feeding subject
* Positive urine pregnancy screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm, Sainte-Foy, Quebec, Canada